CLINICAL TRIAL: NCT05797129
Title: CEDM as a Screening Tool for Breast Cancer in Higher-risk Women: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chen-Pin Chou, Radiologist, Kaohsiung Veterans General Hospital.
Other Study IDs: VGHKS18-CT11-17
Record Dates: First submitted 2023-03-08; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; Contrast-enhanced digital mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CEDM — Women underwent CEDM screening

SUMMARY:
To evaluate the effectiveness of Contrast-enhanced digital mammography (CEDM) in detecting breast cancer in women at higher risk.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effectiveness of different imaging techniques for detecting breast cancer in women with a higher risk due to personal or family history of the disease.

ELIGIBILITY:
Inclusion Criteria:

* women underwent CEDM screening

Exclusion Criteria:

* incomplete imaging exams

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women underwent CEDM screening at Kaohsiung Veterans General Hospital from January 2019 to December 2021
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of cases received and diagnosed with breast cancer (Number) | Up to 3 years
  This refers to the total number of individuals who underwent breast cancer screening or assessment and the number diagnosed with breast cancer. Evaluating the accuracy of screening tests using measures such as true positives and true negatives is crucial for assessing the reliability of screening tests and identifying potential issues. These measures help healthcare professionals make informed decisions about screening and diagnostic strategies.

SECONDARY OUTCOMES:
Total number of cases received and diagnosed as positive requiring a biopsy and MRI (Number) | Up to 3 years
  This refers to the total number of individuals who underwent breast cancer screening or assessment and tested positive, requiring a biopsy and MRI for further evaluation. A biopsy is necessary to confirm whether an individual has breast cancer. Monitoring the diagnostic accuracy of breast cancer screening tests and the number of individuals requiring further procedures is essential for determining appropriate treatment or monitoring. Measures such as true positives and true negatives are used to evaluate the accuracy of screening tests.
True positive results obtained by the diagnostic method (Number) | Up to 3 years
  The total number of true positive results obtained by the diagnostic method, indicating the cases with breast cancer that are correctly identified. A higher number of true positives demonstrates better performance in correctly identifying cases with breast cancer.
True negative results obtained by the diagnostic method (Number) | Up to 3 years
  The total number of true negative results obtained by the diagnostic method, indicating the cases without breast cancer that are correctly identified. A higher number of true negatives demonstrates better performance in correctly identifying cases without breast cancer and reducing false positives.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Pin Chou, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on reasonable request from the corresponding author. Some data are not publicly available due to their containing information that could compromise the privacy of research participants.